CLINICAL TRIAL: NCT01466543
Title: Effect of Zydena (Udenafil) on Cerebral Blood Flow and Peripheral Blood Viscosity in Normal and Subcortical Vascular Cognitive Impairment Subjects
Brief Title: Effect of Zydena (Udenafil) on Cerebral Blood Flow and Peripheral Blood Viscosity
Acronym: SMCZN01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Duk Lyul Na, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC 2011-05-042
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Vascular Dementia; Subcortical Vascular Dementia
Keywords: Vascular dementia; Subcortical vascular dementia; Phosphodiesterase 5; Udenafil
MeSH Terms: conditions — Dementia, Vascular | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zydena (Udenafil) (Active Comparator): Zydena (Udenafil) 100 mg, once
  Interventions: Drug: Zydena (Udenafil)
- Placebo (Placebo Comparator): placebo medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zydena (Udenafil) — Zydena (Udenafil) 100 mg, one time
  Other Names: Zydena; Udenafil
  Arms: Zydena (Udenafil)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Zydena (Udenafil) has effect on cerebral blood flow and peripheral blood viscosity in normal and subcortical vascular cognitive impairment subjects.

DETAILED DESCRIPTION:
Udenafil is a newly developed selective phosphodiesterase type 5 inhibitor (PDE5i). Since PDE5i is known to relax smooth muscle cells, it is suggested that PDE5i may dilate cerebral vessels and lead to an increase in cerebral blood flow. The main mechanism of subcortical vascular cognitive impairment are hypoperfusion of the brain. Therefore, in this study, the investigators will investigate whether Udenafil can increase cerebral blood flow and also lower peripheral blood viscosity in normal and subcortical vascular cognitive impairment subjects.

ELIGIBILITY:
Inclusion Criteria:

for Normal control group

* Normal cognition by detailed neuropsychological tests
* Brain MRI scan with no or minimal white matter hyperintensities

for Subcortical vascular mild cognitive impairment (svMCI)

* Clinical diagnosis of svMCI
* Brain MRI scan with severe white matter hyperintensities

Exclusion Criteria:

- Contraindications to phosphodiesterase type 5 (Zydena, Udenafil)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | One hour after the administration of the medication
  Measured by Near-infrared spectroscopy (NIRS)

SECONDARY OUTCOMES:
Peripheral blood viscosity | One hour after the administration of the medication
  Measured from whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, MD. PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea